CLINICAL TRIAL: NCT00337506
Title: A Multicenter Open-Label Phase II Study of Velcade Combined With High-Dose Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Velcade Combined With High-Dose Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD 03/6-E
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Last update posted 2006-06-16 (Estimated); Status verified 2004-08

CONDITIONS: Multiple Myeloma
Keywords: the efficacy and safety of Velcade plus dexamethasone; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Bortezomib

INTERVENTIONS:
Drug: Dexamethasone
Drug: velcade

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of Velcade plus dexamethasone used as induction chemotherapy prior to autologous transplantation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MM according to the SWOG criteria (annex 1)
* previously untreated (localized radiotherapy is allowed)
* symptomatic MM stage II or III according to Durie-Salmon staging system (annex 2) or stage I with one symptomatic osteolytic lesion
* with measurable levels of paraprotein in the serum (> 1g/dl) or in the urine (> 0.2g/24h)
* age < 75 years
* able to understand and to given an informed consent
* male, female without childbearing potential or negative urine pregnancy test within 72 hours prior to beginning the treatment. Women of childbearing potential must be following adequate contraceptive measures.
* no active systemic infection. In the presence of any active systemic infection, adequate broad-spectrum or organism-specific antibiotic coverage must be administered. Patients must be a febrile with stable vital signs while receiving antibiotics for at least 48 hours prior to beginning the treatment with Velcade plus dexamethasone.

Exclusion Criteria:

* life expectancy < 2 months
* ECOG performance status > 2 (annex 3)
* proven amyloidosis
* positive HIV serology
* antecedents of severe psychiatric disease
* severe diabetes contraindicating the use of high-dose corticoïds
* > NCI grade 2 peripheral neuropathy (Annex IV)
* serum biochemical values as follow

  * creatinin level > 200mmol/l
  * bilirubin, transaminases or gGT > 3 the upper normal limit
* use of any experimental drugs within 30 days of baseline

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-08

PRIMARY OUTCOMES:
Complete remission after 4 cycles:
disappearance of serum and/or urine M-component (confirmed by immunofixation)
< 5% plasma cells in the bone marrow resolution of all extra-osseous plasmacytomas
no evidence of bone progression

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc HAROUSSEAU, MD, Principal Investigator — NANTES UH
Locations (1):
- Jean-Luc HAROUSSEAU, Nantes, France